CLINICAL TRIAL: NCT06622850
Title: Effect of Acupressure on Pain, Anxiety and Hemodynamic Variables in Patients Undergoing Urodynamics: A Randomized Controlled Study
Brief Title: Effect of Acupressure on Pain, Anxiety and Hemodynamic Variables in Patients Undergoing Urodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Assistant Professor, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TU-BOZKUL-009
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Pain; Acupressure; Urodynamics
Keywords: Urodynamics; Pain; Anxiety; Acupressure
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-arm (1:1), randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: During the data collection process, patients will be assessed for inclusion in the study by the researcher M.B. when the patients come to the urology outpatient clinic. Block randomization will be applied to eliminate selection bias. Patients will be assigned to acupressure and placebo acupressure groups according to the permutations (ABBAAB, BABABA, etc.) in the randomization list created in the computer environment by the biostatistician who is not involved in the study. After the randomization list is created, the representation of group A and B to the experimental or control group will be determined by lottery. M.B., who will not be involved in the data collection process of the study, will write numbers from 1 to 68 on the envelope as many as the number of the sample and the letter A or B representing the groups will be added inside the envelopes. M.B. will open the numbered envelope and inform GB which group the patient is in. All other researchers other than M.B. will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupressure group (Experimental): In acupressure, "cun" is used as the unit of measurement to determine the points to be applied. In order to find the acupressure points correctly, measurements should be made using the individual's own fingers. The thumb widths of the individuals participating in the study will be measured and converted as centimeter 1 cun unit. The points to be used in acupressure will be Shen Men (HT7) located in the transverse wrist crease, in the small depression between the pisiform and ulna bones, (LI11) located at the end of the crease when the elbow is bent, and Hegu (LI4) located in the space between the thumb and index finger will be marked by the certified researcher (GB) with an acetate pen in the patients in the study group. And the application will be performed by the certified researcher (GB).
  Interventions: Other: Acupressure
- Control group (No Intervention): The control group will receive routine care.

INTERVENTIONS:
Other: Acupressure — In acupressure, "cun" is used as the unit of measurement to determine the points to be applied. In order to find the acupressure points correctly, measurements should be made using the individual's own fingers. The thumb widths of the individuals participating in the study will be measured and converted as centimeter 1 cun unit. The points to be used in acupressure will be Shen Men (HT7) located in the transverse wrist crease, in the small depression between the pisiform and ulna bones, (LI11) located at the end of the crease when the elbow is bent, and Hegu (LI4) located in the space between the thumb and index finger will be marked by the certified researcher (GB) with an acetate pen in the patients in the study group. And the application will be performed by the certified researcher (GB).
  Arms: Acupressure group

SUMMARY:
The study was planned as a randomized controlled experimental study to determine the effect of acupressure on pain, anxiety and hemodynamic variables in patients undergoing urodynamics. The study conducted by Azarkhavarani et al. (2024) to determine the effect of acupressure on pain in elderly female patients undergoing extracorporeal shock wave lithotripsy was used as a reference in the calculation of sample size. In the study, the effect size of the difference between pain intensity after acupressure (6.33 ± 0.54 in the experimental group and 7.36 ± 0.54 in the control group) was calculated as Cohen's d: 1,907. In order to reach a higher sample size, the minimum sample size was calculated as 34 in each group in the G*Power (3.1) program with d=0.8, (1- α, bidirectional), 90% power, taking the large effect size limit of 0.8 as a reference. Descriptive Information Form, Visual Analog Scale, State Anxiety Scale and Hemodynamic Variables Monitoring Form will be used to collect the research data. After the forms are applied to the patients and recorded, it will be determined whether they will be in the study or control group according to the randomization schedule. Acupressure will be applied to the patients in the study group by a certified researcher who has completed acupressure courses. The control group will receive routine care. After the acupressure application is completed, urodynamics will be performed. Pain, anxiety levels and hemodynamic variables will be re-evaluated immediately and 15 minutes after the procedure. The data obtained in the study will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 25.0 program. Descriptive statistical methods will be used to evaluate the data. Parametric nonparametric tests will be used according to the suitability of the data used for normal distribution.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled experimental study to determine the effect of acupressure on pain, anxiety and hemodynamic variables in patients undergoing urodynamics. The study conducted by Azarkhavarani et al. (2024) to determine the effect of acupressure on pain in elderly female patients undergoing extracorporeal shock wave lithotripsy was used as a reference in the calculation of sample size. In the study, the effect size of the difference between pain intensity after acupressure (6.33 ± 0.54 in the experimental group and 7.36 ± 0.54 in the control group) was calculated as Cohen's d: 1,907. In order to reach a higher sample size, the minimum sample size was calculated as 34 in each group in the G*Power (3.1) program with d=0.8, (1- α, bidirectional), 90% power, taking the large effect size limit of 0.8 as a reference. Descriptive Information Form, Visual Analog Scale, State Anxiety Scale and Hemodynamic Variables Monitoring Form will be used to collect the research data. After the forms are applied to the patients and recorded, it will be determined whether they will be in the study or control group according to the randomization schedule. Acupressure will be applied to the patients in the study group by a certified researcher who has completed acupressure courses.The points to be used in acupressure will be Shen Men (HT7) located in the transverse wrist bend, in the small depression between the pisiform and ulna bones, (LI11) located at the end of the bend when the elbow is in the bent position, and Hegu (LI4) located in the space between the thumb and index finger will be marked by the certified researcher (GB) with an acetate pen in the patients in the study group. And the application will be performed by the certified researcher (GB). Patients in the control group will not receive any application and will receive routine care. After the acupressure application is completed, urodynamics will be performed. Pain, anxiety levels and hemodynamic variables will be re-evaluated immediately and 15 minutes after the procedure. The data obtained in the study will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 25.0 program. Descriptive statistical methods will be used to evaluate the data. Parametric nonparametric tests will be used according to the suitability of the data used for normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the study,
* 18 years of age or older,
* Conscious, oriented and cooperative,
* No communication problems,
* Individuals undergoing invasive urodynamic procedures.

Exclusion Criteria:

* Who did not agree to participate in the study,
* Under 18,
* Conscious, oriented and uncooperative,
* Communication problems,
* Individuals who did not undergo invasive urodynamics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Pain score | 10 months
  Visual Analog Scale: It is a scale that provides a subjective assessment of pain on a horizontal or vertical line from 0 (no pain at all)-10 (very severe pain) to evaluate the level of pain (Wewers and Lowe, 1990).
Anxiety | 10 months
  The State Anxiety Scale : In this study, the DAQ, which is structured to measure momentary feelings, was used. Its Turkish validity and reliability was conducted by Öner and Le Compte in 1983. The DAQ consists of 20 questions on a four-point Likert scale. The statements in the DAQ are evaluated as not at all (1), a little (2), a lot (3) and completely (4). In this section, the statements are divided into direct and reversed statements. Inverted statements: 1st, 2nd, 5th, 5th, 8th, 8th, 10th, 11th, 15th, 16th, 19th, 20th items. The total score of the reversed statements is subtracted from the total score of the direct statements and the number 50, which is the invariant value of the DAQ, is added to the value obtained and the DAQ score is calculated. The scale score ranges between 20-80 and an increase in the score indicates an increase in the level of anxiety.
Hemodynamic Variables | 10 months
  Hemodynamic Variables Monitoring Form : In this form, hemodynamic variables of the study and control groups measured before, immediately after and 15 minutes after the procedure will be recorded. Patient values will be measured and recorded by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Uğraş, Principal Investigator — Mersin University; Elife KETTAŞ DÖLEK, Principal Investigator — MERSIN UNIVERSITY HOSPITAL; Murat BOZLU, Principal Investigator — MERSIN UNIVERSITY HOSPITAL; Gamze Bozkul, Study Director — Tarsus Üniversitesi
Locations (1):
- Mersin University, Mersin, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Safdari A, Khazaei S, Biglarkhani M, Mousavibahar SH, Borzou SR. Effect of acupressure on pain intensity and physiological indices in patients undergoing extracorporeal shock wave lithotripsy: a randomized double-blind sham-controlled clinical trial. BMC Complement Med Ther. 2024 Jan 25;24(1):55. doi: 10.1186/s12906-024-04360-1. PMID 38273233
- [Background] Restawan I.G., Sjattar A.L. & Irwan A.M. (2023). Effectiveness of acupressure therapy in lowering blood pressure in patients with hypertension: A systematic review. Clinical Epidemiology and Global Health. 21. https://doi.org/10.1016/j.cegh.2023.101292
- [Background] Monson E, Arney D, Benham B, Bird R, Elias E, Linden K, McCord K, Miller C, Miller T, Ritter L, Waggy D. Beyond Pills: Acupressure Impact on Self-Rated Pain and Anxiety Scores. J Altern Complement Med. 2019 May;25(5):517-521. doi: 10.1089/acm.2018.0422. Epub 2019 Mar 30. PMID 30932686
- [Background] Jiang ZF, Liu G, Sun XX, Zhi N, Li XM, Sun R, Zhang H. Auricular acupressure for constipation in adults: a systematic review and meta-analysis. Front Physiol. 2023 Oct 16;14:1257660. doi: 10.3389/fphys.2023.1257660. eCollection 2023. PMID 37908337
- [Background] Drake MJ, Doumouchtsis SK, Hashim H, Gammie A. Fundamentals of urodynamic practice, based on International Continence Society good urodynamic practices recommendations. Neurourol Urodyn. 2018 Aug;37(S6):S50-S60. doi: 10.1002/nau.23773. PMID 30614058
- [Background] Biardeau X, Lam O, Ba V, Campeau L, Corcos J. Prospective evaluation of anxiety, pain, and embarrassment associated with cystoscopy and urodynamic testing in clinical practice. Can Urol Assoc J. 2017 Mar-Apr;11(3-4):104-110. doi: 10.5489/cuaj.4127. PMID 28515809
- See also: Related Info — https://doi.org/10.1016/j.urology.2020.06.035